CLINICAL TRIAL: NCT05248048
Title: Hepatic Artery Transfusion of NKG2D CAR-T Cells to Treat Patients With Previously Treated Liver Metastatic Colorectal Cancer: a Prospective, Multicenter Clinical Trial
Brief Title: NKG2D CAR-T Cells to Treat Patients With Previously Treated Liver Metastatic Colorectal Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Hangzhou Cheetah Cell Therapeutics Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CART-002
Record Dates: First submitted 2022-02-08; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: Refractory Metastatic Colorectal Cancer; NKG2D; CAR-NK
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunotherapy, Adoptive; NK Cell Lectin-Like Receptor Subfamily K; Automobiles; Cell Count

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NKG2D CAR-NK (Experimental): CAR-T infusion
  Interventions: Biological: CAR-T infusion

INTERVENTIONS:
Biological: CAR-T infusion — NKG2D CAR-NK Cell Therapy in Patients With Refractory Metastatic Colorectal Cancer
  Other Names: Natural killer group 2 member D (NKG2D) ligand-targeting chimeric antigen receptor (CAR) natural killer (NK) cells

SUMMARY:
Evaluate the clinical safety and feasibility of NKG2D CAR-T administrated by hepatic artery transfusion for patients with previously treated liver metastatic colorectal cancer.

DETAILED DESCRIPTION:
Evaluate the clinical safety and feasibility of NKG2D CAR-T administrated by hepatic artery transfusion for patients with previously treated liver metastatic colorectal cancer. Evaluate the maximum tolerated dose (MTD), dose limiting toxicities (DLT), and toxicity spectrum of NKG2D CAR-T treatment administrated by hepatic artery transfusion. Secondary Objectives: Evaluate the efficacy of NKG2D CAR-T administrated by hepatic artery transfusion for patients with previously treated liver metastatic colorectal cancer, including PSF, DCR, SD >= 8 weeks, ORR, OS, and DOR.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to performing any study protocol-related procedures other than routine care, a voluntarily signed and dated subject informed Consent Form (ICF) must be obtained in accordance with regulatory and institutional guidelines.
2. Aged 18-75 years.
3. There is definite histological evidence of adenocarcinoma of the colon or rectum.
4. The Eastern Cooperative Oncology Group (ECOG) performance Status (PS) score was 0-1 (see Appendix 1).
5. Liver metastasis was confirmed by PET-CT, CT, MR, and/or intraoperative exploration (histological diagnosis is not required).
6. According to the response evaluation criteria in solid Tumors (RECIST) (Version 1.1), patients have at least one target lesion with a measurable diameter line (CT scan of tumor lesion length >= 10 mm, The short diameter of CT scan of lymph node lesions >= 15 mm, and the scanning layer thickness is no more than 5 mm).
7. Failure of treatment after previous standard chemotherapy for metastatic colorectal cancer (including disease progression and unacceptable adverse reactions):

(1)Chemotherapy regimens must include fluorouracil (5-fluorouracil/capecitabine /S-1), oxaliplatin and irinotecan (2)Patients receiving oxaliplatin in adjuvant therapy should develop disease progression during adjuvant therapy or within 6 months after completion of adjuvant therapy; (3)patients may have previously received bevacizumab and/or cetuximab and/or rigfinil and/or furoquitinib.

8. The primary tumor of the colon or rectum has been surgically removed, or the liver metastases are considered to be irretrievable after the evaluation of a multidisciplinary colorectal cancer team consisting of at least two gastrointestinal surgeons, one hepatobiliary surgeon, one oncologist, one interventional surgeon, and one radiologist.

9. The following laboratory test values obtained during the root screening period (reaching the standard and stable before participating in the study) have appropriate organ functions: Neutrophil count >= 1.5 x 109/L, platelet count >= 75 x 10^9/L, serum total bilirubin <= upper normal limits UNL), aspartate aminotransferase <= 2 x UNL, alanine aminotransferase <= 2 x UNL, serum creatinine <= 1.5 x UNL.

10. Negative urine or serum pregnancy tests in women of reproductive age within 7 days prior to treatment.

Exclusion Criteria:

1. The presence or co-existence of other active malignancies (other than those that have been curable for more than 5 years and have received curative treatment or carcinoma in situ that can be cured with adequate treatment).
2. Subjects have central nervous system metastasis or previous brain metastases.
3. Had received hepatic arterial infusion chemotherapy, hepatic arterial embolization chemotherapy or hepatic radiotherapy within 3 months.
4. Received liver surgery (except biopsy for liver metastasis) and liver interventional ablation within the previous 3 months.
5. CT angiography showed severe arterial embolism or hepatic arterial variation.
6. Partial prothrombin time (APTT) or prothrombin time (PT) exceeded 1.5 x ULN (based on the normal value in the clinical trial research center), or patients with evidence or history of bleeding tendency within 2 months prior to enrollment, regardless of severity.
7. Active infection less than 7 days after completion of systemic antibiotic therapy.
8. Major surgery or severe trauma, such as laparotomy, thoracotomy, laparoscopic viscerectomy, etc. within 4 weeks prior to enrollment (surgical incisions should be completely healed before randomization).
9. Active coronary artery disease, severe/unstable angina or newly diagnosed angina or myocardial infarction within 12 months prior to enrollment.
10. Thrombosis or embolism events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, and deep vein thrombosis, occurred within 12 months prior to enrollment.

The New York Heart Association (NYHA) has grade II congestive Heart failure or higher (see Appendix 2).

12. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis (hepatitis B, defined as HBV-DNA >= 500 IU/ mL; Hepatitis C, defined as hcV-RNA higher than the lower limit of the assay) or co-infection with hepatitis B and c.

13. Presence of any active, known or suspected autoimmune disease. Subjects who are in a stable state and do not require systemic immunosuppressive therapy, such as type I diabetes, hypothyroidism requiring only hormone replacement therapy, and skin conditions that do not require systemic therapy (e.g., vitiligo, psoriasis, and hair loss) are allowed to be enrolled.

14. Presence of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic disease (e.g., diabetes, hypertension, pulmonary fibrosis and acute pneumonia).

15. Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) grade 2 or above toxicity (except anaemia, hair loss, skin pigmentation) arising from any prior treatment that has not subsided.

16. Programmed death-1 within 3 months Pd-1) or its ligand (PD-L1) antibody, anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4) antibody, or other drugs/antibodies that act on T cell co-stimulation or checkpoint pathways.

17. Positive pregnancy test before first use in women who are pregnant or breast-feeding or who are at risk of pregnancy.

18. The investigator considers that the subject has any clinical or laboratory abnormalities or compliance issues that make it inappropriate to participate in this clinical study.

19. There are serious psychological or mental abnormalities. 20. Participated in clinical trials of other drugs within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity#DLT# | 28 days
  Safety
Maximal Tolerable Dose#MTD# | 28 days
  tolerability evaluation

SECONDARY OUTCOMES:
Antitumor efficacy-Objective response rate (ORR) | 52 weeks
  The number of cases in which tumor size is reduced to partial response (PR) or complete response (CR) / the total number of evaluable cases (%).
Antitumor efficacy-Overall survival (OS) | 52 weeks
  The period from the first study treatment to any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Xuehu Xu, MD, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China